CLINICAL TRIAL: NCT03624998
Title: The Effects of Cognitive and Behavioral Functioning on Gait Rehabilitation in Orthopedic Patients Submitted to Total Hip Arthroplasty
Brief Title: The Effects of Cognitive Functioning on Gait Rehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: L3031
Record Dates: First submitted 2018-05-23; First posted 2018-08-10 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Total Hip Arthroplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- THA Patients (Experimental): Orthopedic patients submitted to elective surgery (THA - Total Hip Arthroplasty)
  Interventions: Other: Cognitive and physiatric testing

INTERVENTIONS:
Other: Cognitive and physiatric testing — Neuropsychological test battery and physiatric tests

SUMMARY:
The present study is designed to investigate whether the behavioral and cognitive functioning might predict the outcome of the rehabilitation of gait related abilities in orthopedic patients submitted to elective surgery (total hip arthroplasty). The evaluation of gait related abilities will be performed with specific physiatric tests, while cognitive functioning will be studied by means of an extended neuropsychological battery.

ELIGIBILITY:
Inclusion Criteria:

* Age comprised between 50 and 80 years
* Submission to total hip arthroplasty
* Admission to the local rehabilitation program
* Signature of the informed consent

Exclusion Criteria:

* Major medical issues (e.g. neurologial or neurodegenerative diseases)
* Assumption of psychiatric drugs
* Pregnancy

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-04-03 (Actual); Primary Completion 2020-04-02 (Estimated); Study Completion 2020-04-02 (Estimated)

PRIMARY OUTCOMES:
Relationship between the cognitive functioning and gait rehabilitation | The first measures will be taken at the enrollment, at 7 days after the enrollment and at 15 days after the enrollment.
  We will measure the patients' cognitive functioning, investigated by means of a extensive neuropsychological and behavioral battery and the outcome of gait rehabilitation, measured at the enrollment, at 7 days after the enrollment and at 15 days after the enrollment.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Galeazzi, Milan, Italia, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Negrini F, Preti M, Zirone E, Mazziotti D, Biffi M, Pelosi C, Banfi G, Zapparoli L. The Importance of Cognitive Executive Functions in Gait Recovery After Total Hip Arthroplasty. Arch Phys Med Rehabil. 2020 Apr;101(4):579-586. doi: 10.1016/j.apmr.2019.12.004. Epub 2020 Jan 7. PMID 31917194